CLINICAL TRIAL: NCT01535716
Title: Does Goal-directed Hemodynamic Therapy Driven by Endotracheal Cardiac Output Monitoring System During Surgical Intervention Reduce Hospital Stay and Major Adverse Cardiac Events Following Cardiac Surgery?
Brief Title: Effects of a Goal-directed Hemodynamic Therapy Driven by ECOM on Morbidity and Mortality After Cardiac Surgery?
Acronym: ECOMIII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-A01210-41
Record Dates: First submitted 2012-02-07; First posted 2012-02-20 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Surgery With Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECOM group (Experimental): 50 Patients scheduled for elective coronary surgery with cardiopulmonary bypass
  Interventions: Behavioral: hemodynamic optimization strategy driven by the ECOM
- standard management group (Active Comparator): 50 Patients scheduled for elective coronary surgery with cardiopulmonary bypass
  Interventions: Behavioral: standard management strategy

INTERVENTIONS:
Behavioral: hemodynamic optimization strategy driven by the ECOM — goal directed hemodynamic therapy is based on the ECOM evaluation of stroke volume variation (SVV) & cardiac index (CI).
  goals:
  * SVV < 11%
  * IC > 2,2 ml/min/m²
  During the anesthesia
  Other Names: Endotracheal cardiac output monitoring
  Arms: ECOM group
Behavioral: standard management strategy — goal directed hemodynamic therapy will be set and performed by the attending anesthetist, based on the analysis of further clinical parameters: Standard monitoring : heart rate, saturation index
  * Diuresis > 0,5ml/kg/h
  * Blood pressure , PAM > 65 mmHg
  * Pulse pressure variation
  * CVP 8 to 12 cmH20
  * Visual aspect of the heart
  * Overload signs During the anesthesia
  Arms: standard management group

SUMMARY:
Goal-directed hemodynamic and fluid optimizations are shown to be a key factor of the medical care during anesthesia.According to medical literature, goal-directed fluid and hemodynamic optimizations are more efficient when based on the dynamic parameters than when based on the statics ones, and the major dynamic criteria is the cardiac output. Unfortunately, transpulmonary thermodilution, the device considered as "The gold standard" to evaluate cardiac output is associated with many complications.Furthermore, devices commercialized in the past decade were not able to replace the transpulmonary thermodilution.

As all monitoring devices aren't reliable enough to be widely used in practice they are left aside in benefits of the clinical evaluation. Even though, hemodynamic optimization based on the analysis of several clinical parameters seems to guarantee good cares thanks to a favorable benefits/risks balance, it could be improved by new plug and play mini-invasive systems.

In the investigators opinion, the ECOM system seems able to provide a monitoring tool which responds to all the expectations of a modern hemodynamic monitoring device. It uses a well known technique, the bioimpedance. The investigators suppose this device should be more efficient than the one that has been used before. Indeed, as the system is build on the endotracheal tube, it comes closer to the aorta, where all the measures are made, and the recorded signal should be less affected by the passage through the surrounding tissues.

This randomized and controlled trial will study Patients scheduled for elective coronary surgery with cardiopulmonary bypass.

The purpose of this trial is to evaluate the benefits of an intraoperative goal-directed hemodynamic therapy based on the ECOM cardiac output measure on mortality and major postoperative cardiac morbidity after coronary surgery, when compared with a standard management strategy.

Patients will be allocated into control and ECOM groups, of 50 peoples each. The standard management strategy, applied to the control group, will be set and led by the attending anesthetist, based on the analysis of further clinical parameters. The ECOM Group will face the hemodynamic optimization strategy led by the ECOM evaluation of cardiac output and stroke volume variation.

The main hypothesis is that the hemodynamic strategy led by the ECOM cardiac output measure will reduce mortality and morbidity after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any man or woman
* Over 18 year-old
* After obtaining written informed consent
* Scheduled for elective coronary surgery with CPB

Exclusion Criteria:

* Emergency surgery (< 24h)
* Combined cardiac surgery
* Patients < 18 years-old and/or unable to give informed consent
* Patients who refuse to give informed consent
* Pregnancy
* PVC allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | Data collected at the exit of hospital or at death, if during hospital stay.patients will be followed for the duration of hospital stay, an expected average of 10 days. expected before 1 month

SECONDARY OUTCOMES:
Number of major adverse cardiac events during stay in hospital | Data collected at the exit of ICU, at the exit of hospital or at death if during hospital stay.patients will be followed for the duration of hospital stay, an expected average of 10 days.Up to 1 month
Length of stay in ICU | at the exit of ICU or at death, if during hospital stay.expected before 1 month
In-hospital mortality | at the end of the study. up to 12 month
Number of patients with Major adverse cardiac events during in-hospital stay. | at the end of the study. Up to 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Fellahi, Study Director — EA3212: groupe coeur et ischémie
Locations (1):
- University Hospital of Caen, Caen, Calvados, France